CLINICAL TRIAL: NCT06552273
Title: Implementation of a Self-applied Online Psychological Intervention for Emotional Reasoning Bias in People With Public Speaking Anxiety: A Randomized Controlled Trial
Brief Title: Online Psychotherapy for Emotional Reasoning Bias in Public Speaking Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Macarena Paredes Mealla, PhD Student, Universitat Jaume I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEISH/86/2023
Record Dates: First submitted 2024-07-11; First posted 2024-08-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Public Speaking Anxiety
Keywords: Bias correction training; Emotional reasoning; Public speaking anxiety; Internet intervention; Self-applied intervention; Randomized controlled trial; Scared of speaking in public; Transdiagnostic process; Social anxiety

STUDY DESIGN:
Intervention Model Description: Two arms are compared, an experimental group to which bias correction training will be applied and a control group, to which a non-specific mindfulness intervention will be used. Subjects will be randomly assigned to one group or the other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Reasoning bias correction training (Experimental): The experimental arm will receive an Emotional Reasoning bias correction training. The training consists of 12 self-administrated sessions, delivered online.
  Interventions: Behavioral: Emotional Reasoning bias correction training
- Intervention based on mindfulness (Active Comparator): The control group refers to an intervention based on mindfulness skills. This treatment is part of a Transdiagnostic treatment developed in our laboratory, for the treatment of patients with emotional disorders (Díaz-García et al., 2017).
  Interventions: Behavioral: Module of Mindfulness of the Transdiagnostic treatment

INTERVENTIONS:
Behavioral: Emotional Reasoning bias correction training — Emotional Reasoning Bias correction training involves 12 daily self-applied sessions focusing on psychoeducation about emotions and identifying ER biases and their impact on behaviour.
  Arms: Emotional Reasoning bias correction training
Behavioral: Module of Mindfulness of the Transdiagnostic treatment — Module based on mindfulness using techniques for training in awareness and acceptance of experiences, observing experiences as they arise without judgment.
  Arms: Intervention based on mindfulness

SUMMARY:
The study aims to develop and implement a self-applied online psychological intervention for the correction of Emotional Reasoning bias for people with public speaking anxiety. By comparing the effects of this training for ER biases vs. a non-specific mindfulness intervention, the newly developed intervention is expected to promote a greater reduction in emotional reasoning bias and the severity of symptomatology associated with public speaking anxiety.

DETAILED DESCRIPTION:
Among anxiety disorders, one of the most common is Social Anxiety Disorder. Particularly, the specific subtype performance only, i.e., public speaking anxiety, has a prevalence rate of 33% in community samples, being one of the disorders that cause major occupational, educational and social interferences, which represent a high impact on daily functioning. Several cognitive factors may prevent patients from correcting negative thinking; one is the Emotional Reasoning bias. Therefore, in the present study, the aim is to implement training for correcting Emotional Reasoning biases as a transdiagnostic process in people with public speaking anxiety. Regarding implementation and dissemination, it is proposed that this treatment be Internet-based and delivered through information and communication technologies (ICT).

To evaluate the effects of this intervention, a randomized controlled trial will be conducted, comparing two arms, an experimental group to which the bias correction training will be applied and a control group, to which a non-specific intervention will be used. A total of 158 participants based on calculations with the G*Power program will be randomly allocated to an intervention group (N=79) and a control group (N=79). Bias correction training consists of 12 daily self-applied sessions in which components such as psychoeducation in emotions and the detection of ER biases and their impact on behavior are targeted. The primary outcome measure will be Emotional reasoning bias severity and symptomatology associated with public speaking anxiety. Secondary outcome measures will be the severity of depressive and anxious symptomatology, quality of life, usability, and perceived acceptance of participants.

Individuals will be assessed thrice: at baseline, post-treatment, and 3-month follow-up.

Data will be analyzed both per protocol and intention-to-treat. This study will pioneer this type of intervention by bringing together an underdeveloped concept with implementing new technologies. It is intended to increase our knowledge about treatments administered through the Internet and will contribute to improving the dissemination of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Be of legal age.
2. Accept the informed consent.
3. Adequately understand/read Spanish.
4. Have access to a mobile device or computer with an Internet connection.
5. Not receiving any other psychological treatment for public speaking anxiety during the study period.
6. Have a score of 43 or higher on the Emotional reasoning scale (ERPSAS) AND a score of 55 or higher on the Spanish version of the Public Speaking Anxiety Scale (PSAS-S) for fear of public speaking.
7. If taking prescribed medication for anxiety/depression, have had no changes in dosage for at least one month before the procedure.

Exclusion Criteria:

1. Not accepting the informed consent.
2. Being a minor.
3. Having a severe mental disorder (bipolar disorder, schizophrenia, or other psychotic disorders) or substance abuse (alcohol or other substances) or having active suicidal plans (suicide item in the ODSIS depression questionnaire ≥ 2) that would prevent participation in the program.
4. In the case of receiving medication, changes in medication during treatment will be evaluated but will not lead to exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ERPSAS Emotional Reasoning Public Speaking Anxiety Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 13th day (Post-treatment evaluation) and 3-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 3 month follow-up.
  ERPSAS is a self-report instrument consisting of the presentation of 4 scenarios with different endings depending on whether objective safety or danger information is presented and whether there is an anxiety response or not. Based on these scenarios the participant must measure, on a visual analog scale (VAS) from 0 to 100, the degree of danger, safety, controllability, desire to avoid the situation and degree of discomfort. The sum of these scales provides a single perceived threat score providing a measure to determine the presence of the Emotional Reasoning Bias. If the participant evaluates emotional situations as threatening without objective information of danger, the presence of an Emotional Reasoning bias arises. The scale has a range of 0-96 points (M= 36.57; SD= 14.18). The higher the score, the greater the emotional reasoning bias, with the cut-off point being a score of 47. Participants scoring above half a standard deviation above the mean will be included.
Changes in Public Speaking Anxiety Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 13th day (Post-treatment evaluation) and 3-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 3 month follow-up.
  The Public Speaking Anxiety Scale, which contains 17 items with a 5-point Likert-type response format (1=Not at all, 5=Extremely). This scale measures the presence and severity of cognitive, behavioural, and physiological symptomatology related to fear of public speaking, with a cut-off point of 73 (M= 49.33; SD= 12.88). Participants scoring above half a standard deviation above the mean will be included.

SECONDARY OUTCOMES:
Changes in Overall Anxiety Severity and Impairment Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 13th day (Post-treatment evaluation) and 3-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 3 month follow-up.
  OASIS is a 5-item self-report instrument that assesses a unidimensional factor related to the severity and frequency of anxiety symptoms, as well as behavioral avoidance and functional impairment associated with these symptoms in the past week. Each item has five response options, coded from 0 to 4. The total score is calculated by adding the values of all items, ranging from 0 to 20. Scores higher than 8 indicate the presence of anxiety symptoms. This scale has been validated online in a sample of patients with depression and anxiety, demonstrating good internal consistency (α=0.86), as well as adequate convergent and discriminant validities, and sensitivity to change.
Changes in Overall Depression Severity and Impairment Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 13th day (Post-treatment evaluation) and 3-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 3 month follow-up.
  ODSIS is a 5-item self-report instrument that the severity and functional impairment linked to depression over the past week. Each item has five response options coded from 0 to 4. The total score is calculated by summing the values of all items, ranging from 0 to 20. Scores of 5 or above suggest depressive symptoms. This scale was validated online using a sample of patients with depressive or anxiety disorders. It demonstrates excellent internal consistency (α=0.92), and its construct, convergent, and discriminant validities are supported.
Changes in Quality Life Index | 3 evaluations: at baseline before treatment onset, at treatment completion on the 13th day(Post-treatment evaluation) and 3-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 3 month follow-up.
  The QLI is a 10-item self-report instrument that assesses a single concept of quality of life across 10 dimensions using a ten-point Likert scale (1=poor; 10=excellent). The dimensions include physical well-being, psychological/emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social-emotional support, community and services support, personal fulfillment, spiritual fulfillment, and overall perception of quality of life. The total score is the average of the item scores, ranging from 1 to 10 (1-4.5 = below average quality of life; 4.6-8.1 = average quality of life; 8.2-10 = above average quality of life). The QLI demonstrates high internal consistency (α=0.89) and test-retest reliability (0.89), with discriminant validity evidenced in a sample of psychiatric patients.
Score in System Usability Scale | 2 evaluations: at post-treatment (just after treatment completion on the 13th day) and at 3-month follow up.
  The SUS is a 10-item self-report instrument designed to assess opinions on system usability using a 5-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). The content validity index of the Spanish version of the SUS was favorable, with a rating of 0.92 for item relevance. The Cronbach's α was 0.812.
Score in Satisfaction and acceptance with the training | 2 evaluations: at post-treatment (just after treatment completion on the 13th day) and at 3-month follow up.
  Satisfaction and acceptance with the training will be assessed using questions developed by our team and previously used in studies with technology (Suso-Ribera, Castilla, Zaragozá, Ribera-Canudas, Botella, & García-Palacios, 2018). Examples of items include "To what extent are you satisfied with the intervention?" and "To what extent would you recommend the intervention?".

CONTACTS AND LOCATIONS:
Overall Officials: Macarena Paredes Mealla, PhD Student, Principal Investigator — Universitat Jaume I; Carlos Suso Ribera, Dr., Study Director — Universitat Jaume I; Azucena García Palacios, Dr., Study Director — Universitat Jaume I

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers.

REFERENCES:
- [Background] Diaz-Garcia A, Gonzalez-Robles A, Fernandez-Alvarez J, Garcia-Palacios A, Banos RM, Botella C. Efficacy of a Transdiagnostic internet-based treatment for emotional disorders with a specific component to address positive affect: Study protocol for a randomized controlled trial. BMC Psychiatry. 2017 Apr 20;17(1):145. doi: 10.1186/s12888-017-1297-z. PMID 28424068
- [Background] Paredes-Mealla M, Martinez-Borba V, Miragall M, Garcia-Palacios A, Banos RM, Suso-Ribera C. Is there evidence that emotional reasoning processing underlies emotional disorders in adults? A systematic review. Curr Psychol. 2022 Nov 9:1-17. doi: 10.1007/s12144-022-03884-4. Online ahead of print. PMID 36406838
- [Background] Arntz A, Rauner M, van den Hout M. "If I feel anxious, there must be danger": ex-consequentia reasoning in inferring danger in anxiety disorders. Behav Res Ther. 1995 Nov;33(8):917-25. doi: 10.1016/0005-7967(95)00032-s. PMID 7487851
- [Background] Lommen MJ, Engelhard IM, van den Hout MA, Arntz A. Reducing emotional reasoning: an experimental manipulation in individuals with fear of spiders. Cogn Emot. 2013;27(8):1504-12. doi: 10.1080/02699931.2013.795482. Epub 2013 May 16. PMID 23679871